CLINICAL TRIAL: NCT01330953
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2928057 in Healthy Subjects
Brief Title: A First Human Study of a Ferroportin Antibody
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14151; I5M-FW-FABA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-03-15; First posted 2011-04-07 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
Keywords: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Single intravenous placebo dose.
  Interventions: Drug: Placebo
- 30 mg LY2928057 (Cohort 1) (Experimental): Day 1: single 30-milligram (mg) LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 30-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 30-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 30 mg LY2928057.
  Interventions: Drug: LY2928057
- 100 mg LY2928057 (Cohort 2) (Experimental): Day 1: single 100-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 100-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 100-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 100 mg LY2928057.
  Interventions: Drug: LY2928057
- 300 mg LY2928057 (Cohort 3) (Experimental): Day 1: single 300-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 300-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 300-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 300 mg LY2928057.
  Interventions: Drug: LY2928057
- 1000 mg LY2928057 (Cohort 4) (Experimental): Day 1: single 1000-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 1000-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 1000-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 1000 mg LY2928057.
  Interventions: Drug: LY2928057

INTERVENTIONS:
Drug: Placebo — Single intravenous placebo dose.
  Arms: Placebo
Drug: LY2928057 — Single intravenous dose.
  Other Names: Ferroportin antibody
  Arms: 100 mg LY2928057 (Cohort 2); 1000 mg LY2928057 (Cohort 4); 30 mg LY2928057 (Cohort 1); 300 mg LY2928057 (Cohort 3)

SUMMARY:
The purposes of this study are to evaluate the following in healthy participants: 1) LY2928057 safety, including any side effects possibly associated with LY2928057; 2) how the body processes LY2928057; 3) effect of LY2928057 on blood iron levels; and 4) immune system reactions to LY2928057.

ELIGIBILITY:
Inclusion Criteria:

* Must either be a healthy male (and willing to use reliable birth control method during the study and for 3 months following last study drug dose), or a healthy female who cannot become pregnant
* Must have a body mass index (BMI) between 18.5 and 32.0 kilograms per square meter (kg/m^2), inclusive, and a minimum body weight of 55 kg
* Must have acceptable blood and urine laboratory test results for the study
* Must have suitable veins suitable for easy blood collection and study drug administration
* Must be reliable, follow study procedures, and willing to be available for the duration of the study
* Must have given written informed consent
* Must have acceptable blood pressure and pulse rate for the study

Exclusion Criteria:

* Blood test shows that participant has anemia due to lack of iron
* Currently participating in another clinical study or has completed one less than 30 days ago
* Allergic to biologic agents
* Have previously taken part in this study
* Have abnormal electrocardiogram (ECG) findings that suggest an increased risk with study participation
* Have a history of significant disease that may affect drug actions or pose risk when taking study medication
* Have a history of drug or alcohol abuse
* Are infected with human immunodeficiency virus (HIV)
* Have hepatitis B
* Are pregnant or breastfeeding
* Intend to use over-the-counter or prescription medication within 14 days before dosing, other than oestrogen/progesterone as hormone replacement therapy (HRT). Participants taking these medications are expected to be on chronic, stable doses. Certain medications (for example, vitamin supplements) may be permitted at the discretion of the investigator.
* Have donated more than 450 milliliter (mL) of blood within the last 3 months
* Have a regular alcohol intake greater than 21 units per week (male), or 14 units per week (female), or are unwilling to stop alcohol as required for the study (1 unit = 360 mL of beer, 150 mL of wine, or 45 mL of spirits)
* Are a smoker (smoking more than 10 cigarettes per day) or have used equivalent tobacco products. Participants will not be allowed to smoke while in the study unit.
* Have received live vaccine(s) within 1 month of screening, or intend to during the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) before receiving study drug in this study
* Have a history of atopy, significant allergies to humanized monoclonal antibodies, clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Have any active mental health illness
* Study doctor does not feel the participant should be in the study for any reason

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

REFERENCES:
- [Derived] Sheetz M, Barrington P, Callies S, Berg PH, McColm J, Marbury T, Decker B, Dyas GL, Truhlar SME, Benschop R, Leung D, Berg J, Witcher DR. Targeting the hepcidin-ferroportin pathway in anaemia of chronic kidney disease. Br J Clin Pharmacol. 2019 May;85(5):935-948. doi: 10.1111/bcp.13877. Epub 2019 Mar 4. PMID 30677788

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 mg LY2928057: Day 1: single 30-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 30-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 30-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 30 mg LY2928057.
- 100 mg LY2928057: Day 1: single 100-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 100-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 100-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 100 mg LY2928057.
- 300 mg LY2928057: Day 1: single 300-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: 1 participant receives single 300-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 300-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 300 mg LY2928057.
- 1000 mg LY2928057: Day 1: single 1000-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 1000-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and 7: single 1000-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 1000 mg LY2928057.
Period: Overall Study
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057 | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (13.8) | 33.5 (14.8) | 31.0 (6.3) | 40.2 (11.7) | 27.0 (6.1) | 33.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 0 | 1
  Male | 7 | 6 | 6 | 6 | 6 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 8 | 6 | 6 | 6 | 6 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 8 | 6 | 6 | 6 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Adverse Effects
Description: A clinically significant effect/event was defined as an adverse event (AE). A listing of serious and non-serious AEs is located in the Reported Adverse Event Module.
Time Frame: Baseline through Day 85
Population: The analysis population included all randomized participants dosed with placebo or LY2928057, and who provided safety data at least up to and including the Day 8 assessment.
Measure: Number; unit: participants
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants | 7 | 6 | 5 | 5 | 6

2. Secondary Outcome: Pharmacokinetics, Area Under the Curve (AUC)
Description: Area under the LY2928057 plasma concentration-time curve extrapolated to infinite time (AUC0-∞).
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic AUC analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*h/mL) | 45500 (53) | 1000000 (23) | 4060000 (40) | 19700000 (28)

3. Secondary Outcome: Pharmacokinetics, Maximum Concentration (Cmax)
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic Cmax analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/mL | 4560 (21) | 27400 (14) | 88500 (19) | 276000 (22)

4. Secondary Outcome: Pharmacokinetics, Time to Maximum Concentration (Tmax)
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic tmax analyses.
Measure: Median (Full Range); unit: hour (h)
Groups:
- 30 mg LY2928057: Day 1: single 30-mg LY2928057 intravenous dose; Days 2 and 3: observation period; Days 4 and 5: single 30-mg LY2928057 intravenous dose followed by 24-hour observation period; Days 6 and Day 7: single 30-mg LY2928057 intravenous dose; Days 8-85: participant follow-up for minimum of 12 weeks to assess the safety, immunogenicity, and pharmacokinetic profile of 30 mg LY2928057.
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour (h) | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.50 to 4.00]

5. Secondary Outcome: Pharmacokinetics, Systemic Clearance (CL)
Description: CL=total body clearance of LY2928057 calculated after intravenous administration. Systemic CL was derived from LY2928057 serum concentration data following intravenous administration using classical non compartmental analysis (WinNonlin version 5.3).
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic systemic CL analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
liter per hour (L/h) | 0.6590 (53) | 0.0999 (23) | 0.0739 (40) | 0.0507 (28)

6. Secondary Outcome: Pharmacokinetics, Volume of Distribution (V)
Description: V=LY2928057 steady-state volume of distribution (Vss)
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic Vss analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
L | 13.80 (46) | 4.01 (19) | 3.82 (19) | 4.69 (22)

7. Secondary Outcome: Pharmacokinetics, Terminal Half-Life (t1/2)
Time Frame: Predose, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15, 22, 29, 43, 50, 57, 64, 71, and 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided samples for pharmacokinetic t1/2 analyses.
Measure: Geometric Mean (Full Range); unit: days
Arm/Group | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 6 | 6 | 6 | 6
days | 1.2 [0.9 to 1.5] | 5.1 [3.1 to 7.5] | 6.6 [4.7 to 9.2] | 10.3 [6.1 to 18.0]

8. Secondary Outcome: Change From Baseline in Serum Iron
Description: Maximum change from baseline to any point over 22 days post-infusion.
Time Frame: Baseline, end of infusion, 4, 12, and 24 hours post-infusion on Days 3, 5, 8, 11, 15 and 22
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and provided plasma data for measuring serum iron levels as the primary pharmacodynamic analysis.
Measure: Mean (Standard Deviation); unit: microgram per deciliter (µg/dL)
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
microgram per deciliter (µg/dL) | 32.9 (17.5) | 71.9 (36.1) | 59.9 (22.4) | 95.1 (49.8) | 96.3 (51.9)

9. Secondary Outcome: Number of Participants Forming Antibody to LY2928057
Time Frame: Baseline through Day 85
Population: The analysis population included all randomized participants who received at least 1 dose of LY2928057 and antibody titer results.
Measure: Number; unit: participants
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants | 0 | 3 | 2 | 5 | 4

ADVERSE EVENTS:
Arm/Group | Placebo | 30 mg LY2928057 | 100 mg LY2928057 | 300 mg LY2928057 | 1000 mg LY2928057
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 7/8 | 6/6 | 5/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 30 mg LY2928057 (N=6) | 100 mg LY2928057 (N=6) | 300 mg LY2928057 (N=6) | 1000 mg LY2928057 (N=6)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Catheter site related reaction (General disorders) | 1 (2) | 5 (7) | 3 (5) | 2 (4) | 4 (6)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site erythema (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Infusion site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (4) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes